CLINICAL TRIAL: NCT07399626
Title: Adaptation and Validation of the Hypomanic Personality Scale (HPS-6) to Romanian.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Renata Gheorghiu, Principal Investigator, Babes-Bolyai University
Allocation: Not Applicable | Model: Sequential | Masking: Triple | Purpose: Screening
Other Study IDs: 1068/10.12.2025
Record Dates: First submitted 2026-01-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Bipolar Disorder (BD)
Keywords: bipolar disorder; manic-depression; cyclothymia
MeSH Terms: conditions — Bipolar Disorder; Cyclothymic Disorder

STUDY DESIGN:
Intervention Model Description: The first wave of participants recruits individuals from the community and is meant to pilot the instrument, check its stability and be utilized for exploratory factor analysis. The second wave will be used to test the instrument across DSM-5 validated diagnoses (via SCID-5-CV semi-structured clinical interview) and for confirmatory factor analysis.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Clinical Psychologists conducting the clinical interviews are blinded to participant's diagnosis (from intake form), as well as study scales and scope of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Piloting (Other): Meant for piloting scale, EFA
  Interventions: Diagnostic Test: Hypomanic Personality Scale - 6
- Clinical / Risk Group (Other): Formally clinically evaluated sample, used for CFA
  Interventions: Diagnostic Test: Hypomanic Personality Scale - 6

INTERVENTIONS:
Diagnostic Test: Hypomanic Personality Scale - 6 — A brief instrument, such as the HPS-6, with high specificity can help navigate specialists towards a correct diagnosis or recognize risk patterns in Bipolar Spectrum Individuals.

SUMMARY:
The HPS-6 (Hypomanic Personality Scale, 6 item version) could prove to be a valuable candidate for screening measures of high risk individuals. In the following study, we aim to validate and adapt the HPS-6 for the Romanian population.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a chronic, debilitating disorder, affecting approximately 2.4% of the global population. Inaccurate diagnosis leads to inappropriate management of the disorder as well as unsuitable medication prescription. On average, it can take a BD individual 5 to 10 years to receive an accurate diagnosis and receive competent treatment. Across the European Union (EU) Romania has the lowest prevalence of psychiatric disorders, 14.3%. Unfortunately, these positive estimates are related to the severe stigma linked to poor mental health in the Romanian population. Although the average length of a psychiatric stay in the EU spans across 24.3 days, Romania's average is 17.7. Poor infrastructure and lack of personnel in the Romanian healthcare system might be partially responsible. Therefore, brief, validated screening measures for complex diagnoses are necessary.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Not at high risk of suicide (current)
* Not high SUDs / AUDs (current)
* Native Romanian speaker
* Cognitive abilities intact (reading comprehension of items)

Exclusion Criteria:

* High risk of suicide (current)
* High SUDs / AUDs (current)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Hypomanic Personality Scale - 6 (HPS-6) | Baseline and one month later for re-test measures (in order to account for test-retest reliability)
  The main instrument of the study, the HPS-6 is used to assess bipolar spectrum disorder risk due to and individual's phenotype. The scale contains 6 items and has a binary rating scale ("TRUE" / "FALSE"). The original authors used a cut-off of 3 or higher to represent possible risk for the disorder. Minimum score possible is 0, while the highest is 6.
Mood Disorder Questionnaire (MDQ) | Baseline
  In order to check for convergent validity, the Mood Disorder Questionnaire was administered as well. The instrument screens for a history of manic or hypomanic symptoms. It contains 13 yes or no items created based on the DSM-IV, followed by a 4-point Likert question on the level of impairment; "no problem" to "serious problem" and a 15th item asking is symptoms happened simultaneously. Studies recommend a cut-off of >5 for high risk bipolar populations. The original cut-off of the scale is >7, but it has been criticized for high specificity. The total score is 13 (MIN: 0, MAX: 13).
Behavioral Inhibition System / Behavioral Activation System scales (BISBAS) | One month after Baseline
  The BIS / BAS scales assess two motivational systems, the Behavioral Inhibition System and the Behavioral Activation System. The scale contains 20 items in total. The BAS system, or the approach tendency, is hypothesized to facilitate goal-motivated behavior when presented with incentives, generating an increase in behaviors oriented towards goals, while the BIS motivational system activates inhibition tendencies. Higher scores indicate sensitivity to threats, non-reward (BIS) or the sensitivity towards reward and goal striving (BAS). Total possible score for the BIS subscale is 28 (MIN: 7, MAX: 28), while for the BAS subscale the total possible is 91 (MIN: 13, MAX: 91).
Positive and Negative Affect Schedule (PANAS) | One month after Baseline.
  The Positive and Negative Affect Schedule is a 20-item self-report measure assessing positive and negative affect. Participants rate each item on a 5-point Likert scale ranging from 1 ("very slightly or not at all") to 5 ("extremely"). Each subscale has a possible score range of 10 to 50. Higher PA scores reflect greater energy and concentration, whereas higher NA scores indicate greater levels of distress.
Negative Urgency, Premeditation, Perseverance, Sensations Seeking, and Positive Urgency - Impulsive Behavior Scale (UPPS-P) | One month after Baseline
  The UPPS-P Impulsive Behavior Scale assesses positive and negative emotional urgency along with multiple dimensions of impulsivity. The full instrument includes 59 items across five subscales: Negative Urgency, Positive Urgency, (Lack of) Premeditation, (Lack of) Perseverance, and Sensation Seeking. A scoping review has shown that individuals with bipolar disorder exhibit elevated impulsivity during both positive and negative emotional states, with particularly large effect sizes observed for positive urgency. Because the HPS-6 focuses on positively valenced experiences, only the Positive Urgency subscale was administered in this study. Scores on this subscale range from 14 to 56, with higher average scores indicating greater impulsive tendencies.
Affective Lability Scale - Short Form (ALS-18) | One month after Baseline
  The ALS-18 is an 18-item measure designed to assess shifts between neutral states and intense affect, emphasizing emotional variability rather than current symptom severity. It comprises three main subscales: Anxiety/Depression Shift (5 items), Depression/Elation Shift (8 items), and Anger (5 items). Items are rated on a 4-point Likert scale ranging from 0 ("very uncharacteristic of me") to 3 ("very characteristic of me"). The total raw score ranges from 0 to 54, with higher scores indicating greater affective lability, reflected in more frequent and intense mood shifts.
Positive Overgeneralization (POG) | One month after Baseline.
  The Positive Overgeneralization Scale (POG) measures the "tendency to generalize good experiences in one domain to broader aspects of life". it contains 3 subscales (lateral generalization, upward generalization and social generalization), comprising altogether 16 items. Lower scores represent a higher predisposition towards that type of positive overgeneralization (Subscale 1 - Lateral generalization: MAX - 30, MIN: 6 , Subscale 2 - Upward generalization: MAX - 25, MIN - 5, Subscale 3 - Social generalization: MAX - 25, MIN - 5).
Altman Self-Rating Mania Scale (ASRM) | Baseline
  The instrument evaluates manic symptom presence and their severity using 5 items, rated on a 4-point Likert scale. Total scores span from 0 to 20, and scores of 6 or above suggest a possible presence of hypomanic or manic symptoms.
Food Neophobia Scale (FNS) | Baseline
  The scale measures one's reluctance to try new or unfamiliar foods. The FNS consists of 10 items rated on a 7-point Likert scale. It has been widely used internationally across diverse fields. Five items assess neophobic behavior, defined as fear of new or unfamiliar experiences, while the remaining five assess neophilic behavior, reflecting interest in and enthusiasm for novelty. Higher FNS scores indicate greater levels of neophobia (MIN: 10, MAX: 70).
Patient Health Questionnaire-9 (PHQ-9) | Baseline
  The Patient Health Questionnaire-9 is a diagnostic tool for depression based on DSM-IV criteria. It includes nine items rated on a 4-point Likert scale ranging from 0 ("Not at all") to 3 ("Nearly every day"). Using the algorithm method, a diagnosis is indicated when five or more symptoms have been present for more than half of the days over the past two weeks. Total scores range from 0 to 21. Alternatively, the summed-item approach involves adding the item scores, with a commonly used cutoff of 10 points to indicate major depressive disorder.
Importance of Olfaction (IOS) | Baseline
  The Importance of Olfaction scale assesses core olfactory functions. It consists of 18 items rated on a 5-point Likert scale ranging from 1 ("strongly disagree") to 5 ("strongly agree"). The scale was designed for use across different cultures and age groups. It includes five subscales reflecting various domains of the importance of smell (e.g., mating and bonding). Total scores range from 18 to 90, with higher scores indicating a greater personal importance attributed to the sense of smell.

SECONDARY OUTCOMES:
Psychiatric Diagnostic Screening Questionnaire (PDSQ) | Baseline
  We used 12 of the 13 subscales of the Psychiatric Diagnostic Screening Questionnaire (PDSQ) to screen for additional psychiatric conditions. The depression subscale was excluded because depressive symptoms were assessed separately with the PHQ-9, and participants also underwent a formal clinical evaluation in which depression was examined in greater detail. The PDSQ is a self-administered screening instrument for common mental health disorders. The Romanian version includes 125 items, with higher scores indicating a greater risk for the respective disorder. Using these subscales, we assessed risk for PTSD, bulimia nervosa, obsessive-compulsive disorder, panic disorder, psychosis, agoraphobia, social phobia, alcohol use disorder, medication abuse, generalized anxiety disorder, and hypochondria (health anxiety).
Suicide Behavior Questionnaire-Revised (SBQ-R) | Baseline
  The SBQ-R is a brief, four-item measure that assesses multiple dimensions of suicidality and provides an overall suicide risk score. Scores of 7 or higher indicate elevated risk in non-clinical samples, whereas a cutoff of 8 or higher is used for clinical samples. Participants were not excluded based on suicide risk, as doing so could introduce bias into the research. Total scores range from 3 to 18.

CONTACTS AND LOCATIONS:
Locations (1):
- Babeș-Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Undecided
Ethics regarding the limited clinical sample.

REFERENCES:
- [Background] Wang, H. R., Woo, Y. S., Ahn, H. S., Ahn, I. M., Kim, H. J., & Bahk, W. M. (2015). The validity of the mood disorder questionnaire for screening bipolar disorder: a meta-analysis. Depression and anxiety, 32(7), 527-538. https://doi.org/10.1002/da.22374
- [Background] Kroenke, K., Spitzer, R. L., & Williams, J. B. W. (1999). Patient Health Questionnaire-9 (PHQ-9). APA PsycTests, 10. https://doi.org/10.1037/t06165-000
- [Background] Manea, L., Gilbody, S., & McMillan, D. (2015). A diagnostic meta-analysis of the Patient Health Questionnaire-9 (PHQ-9) algorithm scoring method as a screen for depression. General hospital psychiatry, 37(1), 67-75. https://doi.org/10.1016/j.genhosppsych.2014.09.009
- [Background] Levis, B., Benedetti, A., & Thombs, B. D. (2019). Accuracy of Patient Health Questionnaire-9 (PHQ-9) for screening to detect major depression: individual participant data meta-analysis. bmj, 365. https://doi.org10.1136/bmj.l1476
- [Background] Pliner, P., & Hobden, K. (1992). Development of a scale to measure the trait of food neophobia in humans. Appetite, 19(2), 105-120. https://doi.org/10.1016/0195-6663(92)90014-W
- [Background] Rabadán, A., & Bernabéu, R. (2021). A systematic review of studies using the Food Neophobia Scale: Conclusions from thirty years of studies. Food Quality and Preference, 93, 104241. https://doi.org/10.1016/j.foodqual.2021.104241
- [Background] Sorokowski, P., Sorokowska, A., Misiak, M., & Roberts, S. C. (2023). Developmental changes in food and non-food odor importance-Data from Scotland and Pakistan. Food Quality and Preference, 111, 104963.
- [Background] Meyer, T. D., & Baur, M. (2009). Positive and negative affect in individuals at high and low risk for bipolar disorders. Journal of Individual Differences, 30(3), 169-175.
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Teh, W. L., Si, S. Y., Liu, J., Subramaniam, M., & Ho, R. (2024). The clinical significance of emotional urgency in bipolar disorder: a scoping review. BMC psychology, 12(1), 273.
- [Background] Eisner, L. R., Johnson, S. L., & Carver, C. S. (2008). Cognitive responses to failure and success relate uniquely to bipolar depression versus mania. Journal of Abnormal Psychology, 117(1), 154.
- [Background] Johnson, S. L., Turner, R. J., & Iwata, N. (2003). BIS/BAS levels and psychiatric disorder: An epidemiological study. Journal of psychopathology and behavioral assessment, 25(1), 25-36.
- [Background] Carver, C. S., & White, T. L. (1994). Behavioral inhibition, behavioral activation, and affective responses to impending reward and punishment: the BIS/BAS scales. Journal of personality and social psychology, 67(2), 319.
- [Background] Osman, A., Bagge, C. L., Gutierrez, P. M., Konick, L. C., Kopper, B. A., & Barrios, F. X. (2001). The Suicidal Behaviors Questionnaire-Revised (SBQ-R): validation with clinical and nonclinical samples. Assessment, 8(4), 443-454.
- [Background] Kwapil, T. R., Miller, M. B., Zinser, M. C., Chapman, L. J., Chapman, J., & Eckblad, M. (2000). A longitudinal study of high scorers on the hypomanic personality scale. Journal of Abnormal Psychology, 109(2), 222. https://doi.org/10.1037/0021-843X.109.2.222
- [Background] Schalet, B. D., Durbin, C. E., & Revelle, W. (2011). Multidimensional structure of the Hypomanic Personality Scale. Psychological assessment, 23(2), 504. https://doi.org/10.1037/a0022301
- [Background] Berson, T. R., Sperry, S. H., Walsh, M. A., & Kwapil, T. R. (2022). A critical examination of multidimensionality within the Hypomanic Personality Scale. Comprehensive Psychiatry, 115, 152306. https://doi.org/10.1016/j.comppsych.2022.152306
- [Background] Eckblad, M., & Chapman, L. J. (1986). Development and validation of a scale for hypomanic personality. Journal of abnormal psychology, 95(3), 214. https://doi.org/10.1037//0021-843x.95.3.214
- [Background] Matza, L. S., Rajagopalan, K. S., Thompson, C. L., & De Lissovoy, G. (2005). Misdiagnosed patients with bipolar disorder: comorbidities, treatment patterns, and direct treatment costs. Journal of Clinical Psychiatry, 66(11), 1432-1440. https://doi.org/10.4088/jcp.v66n1114
- [Background] Miller, C. J., Johnson, S. L., Kwapil, T. R., & Carver, C. S. (2011). Three studies on self-report scales to detect bipolar disorder. Journal of affective disorders, 128(3), 199-210. https://doi.org/10.1016/j.jad.2010.07.012
- [Background] Zhong, Y., Chen, Y., Su, X., Wang, M., Li, Q., Shao, Z., & Sun, L. (2024). Global, regional and national burdens of bipolar disorders in adolescents and young adults: a trend analysis from 1990 to 2019. General Psychiatry, 37(1), e101255. https://doi.org/10.1136/gpsych-2023-101255
- [Background] Iovu, M. B., & Breaz, M. A. (2019). The prevalence and burden of mental and substance use disorders in Romania: Findings from the Global Burden of Disease Study 2016. Psychiatria Danubina, 31(4), 457-464. https://doi.org/10.24869/psyd.2019.457
- [Background] Iaru, I., Bucsa, C., Farcas, A., Pop, C., Cristina, A., Armean, S., ... & Mogosan, C. (2023). Utilization of psychotropic medicines in Romania during 1998-2018. Frontiers in Pharmacology, 14, 1157231. https://doi.org/10.3389/fphar.2023.1157231